CLINICAL TRIAL: NCT01162525
Title: Percutaneous Tibial Nerve Stimulation (pTNS) for Patients With Fecal Urge Incontinence
Brief Title: Percutaneous Tibial Nerve Stimulation for Patients With Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Lukas Marti, Attending physician, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pTNS
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Fecal Urge Incontinence; Percutaneous tibial nerve stimulation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pTNS treatment (Experimental)
  Interventions: Procedure: Percutaneous tibial nerve stimulation (pTNS)

INTERVENTIONS:
Procedure: Percutaneous tibial nerve stimulation (pTNS) — A 34 gauge needle in placed close to the tibial nerve about 2-3 cm above the ankle. A self-adhesive surface electrode is placed on the skin. Needle and surface electrode are connected to an electric stimulator and the stimulating current (0 - 10 mA) is increased in 20 steps. When the patient feels a tingling sensation in the foot, stimulating current is set back for one step and the treatment is started (30 min stimulation).
  Other Names: pTNS; peripheral tibial nerve stimulation; peripheral neuromodulation

SUMMARY:
Percutaneous tibial nerve stimulation is introduced as regular treatment option for fecal urge continence at the Cantonal Hospital St. Gallen. During this introduction phase efficiency und adverse events will be monitored in this observational study.

DETAILED DESCRIPTION:
Before treatment patients will have a proctological exam, a proctoscopy, endosonography and anorectal manometry. Incontinence scores (Wexner, Vaizey, Hanley) and quality of life scores (FIQL, VAS) will be recorded.

Treatment consists of 4 phases with decreasing frequency of percutaneous tibial nerve stimulations (pTNS).

During phase 1 weekly stimulations of 30 mins are applied for 12 weeks. After 6 and 12 weeks incontinence scores are recorded. Additionally after the end of phase 1 quality of life is measured and an anorectal manometry is preformed.

Phase 2 lasts for 8 weeks, with 2-3 stimulations/month Phase 3 lasts for 8 weeks, with stimulations every 3 weeks Phase 4 consists of one stimulation in one month.

After phase 4 incontinence scores und quality of life are measured.

ELIGIBILITY:
Inclusion Criteria:

* fecal urge incontinence
* conservative treatment has been performed without success

Exclusion Criteria:

* current anticoagulation treatment
* sphincter defects larger than 120°
* pregnancy
* pace maker
* implanted defibrillators
* severe heart disease
* existing neurological damages
* disposition for strong bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-01; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Fecal Incontinence | 6 weeks
  Jorge Wexner Score (Dis Colon Rectum (1993) 36:77) compared to pretreatment
  * Score for fecal incontinence, with 5 items and score range of 0 - 20
Fecal Incontinence | 12 weeks
  Jorge Wexner Score (Dis Colon Rectum (1993) 36:77) compared to pretreatment
  * Score for fecal incontinence, with 5 items and score range of 0 - 20
Fecal Incontinence | 32 weeks
  Jorge Wexner Score (Dis Colon Rectum (1993) 36:77) compared to pretreatment
  * Score for fecal incontinence, with 5 items and score range of 0 - 20

SECONDARY OUTCOMES:
Fecal Incontinence | before treatment, 6, 12, 32 wks after initial treatment
  Vaizey Score (Gut (1999) 44:77)
  * Fecal incontinence score similar to Wexner Score
Anorectal manometric measurements | 12 weeks
  compared to pre-treatment values
Quality of Life | before treatment, 6, 32 wks after initial treatment
  2 scores for quality of life are measured:
  * Fecal Incontinence Quality of Life (FIQL) (Dis Colon Rectum (2000) 43:9)
  * Visual Analogue Score Patients are asked to score their well-being in respect to the incontinence by marking a horizontal 10 cm line labelled "extremely bad" and "excellent" at both ends
Cost | at the end of the treatment
  total cost of treatment will be evaluated (material, work hours etc)
Adverse Events | for each treatment interval
  adverse events between treatments:
  * pain, bleeding, neurological sensation, other AE
  Adverse events during percutaneous nerve stimulation:
  * pain, bleeding and discomfort
Urinary incontinence | before treatment, 6, 12, 32 wks after initial treatment
  Hanley Score (BMJ (2001) 322:1096)
  * Urinary incontinence score

CONTACTS AND LOCATIONS:
Overall Officials: Lukas T Marti, Dr. med., Principal Investigator — Department of Surgery, Cantonal Hospital St. Gallen
Locations (1):
- Department of Surgery, Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- See also: Website of the Department of Surgery, Cantonal Hospital of St. Gallen (German only) — http://www.chirurgie.kssg.ch/home/unsere_klinik.html